CLINICAL TRIAL: NCT05603234
Title: Evaluating the Effects of Symptom Monitoring on Physical & Emotional Outcomes During Menopause: A Pilot Randomised Controlled Trial
Brief Title: Symptom Monitoring and Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21059
Record Dates: First submitted 2022-10-10; First posted 2022-11-02 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Menopause
Keywords: Menopause; Hot flushes; Women's Health; Symptom Monitoring
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Monitoring Intervention (Experimental): This group reported their symptoms every day for 14 days.
  Interventions: Behavioral: Symptom Monitoring
- Control (No Intervention): This group did not monitor their symptoms every day for the 14 day period, however they did report their symptoms at the beginning and end of the 14 day period

INTERVENTIONS:
Behavioral: Symptom Monitoring — Reporting symptoms each day via a symptom questionnaire
  Arms: Symptom Monitoring Intervention

SUMMARY:
A recent systematic review suggested that symptom monitoring can result in reductions in menopausal symptoms and improvements in health-related behaviours. To date, no studies have experimentally investigated whether symptom monitoring could be beneficial as an intervention for menopausal women.

One hundred menopausal women were randomised into either a Monitoring-intervention or Control group. A mixed between/ within design was employed, with group membership (i.e., Monitoring-intervention or Control) as the between-subjects component, and time (i.e., baseline and 2-weeks follow-up) as the within-subjects component. Dependent variables included symptom reductions and emotional reactions. Secondary outcomes included help-seeking, communication, medical decision-making, health awareness, self-efficacy, and health anxiety.

ELIGIBILITY:
Inclusion criteria:

* Women
* Aged 18+
* Reporting at least 2 menopausal hot flushes per day
* Self-reported peri- or post-menopausal status.

Exclusion criteria:

* Male
* Under age 18
* Reported fewer than 2 hot flushes per day
* Does not self-report peri- or post-menopausal status.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be women experiencing self-reported menopause/ perimenopause
Enrollment: 112 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Menopausal symptom changes via the Daily Record Keeping (DRK) form | at baseline and after 2 weeks of symptom monitoring
  Changes in menopausal symptom scores after 2-weeks of symptom monitoring, where reductions in symptoms would suggest a beneficial outcomes.
Emotional outcomes via the Daily Record Keeping (DRK) form | at baseline and after 2 weeks of symptom monitoring
  Changes in emotion scores after 2-weeks of symptom monitoring. The DRK assesses emotional outcomes via specific emotion subscales including Negative Emotions, Positive affect, Anxiety, Depression, Loneliness. Reductions in Negative Emotions, Anxiety, Loneliness, Depression after 2-weeks would suggest benefical effects, as would increases in Positive Affect.

SECONDARY OUTCOMES:
Help seeking intentions | at baseline and after 2 weeks of symptom monitoring
  Changes in Help Seeking Intention scores as assessed via the General Help Seeking Questionnaire (GHSQ). Increases in GHSQ scores at 2-weeks would indicate benefical effects on help seeking behaviour.
General Self Efficacy | at baseline and after 2 weeks of symptom monitoring
  Changes in General Self Efficacy scores as assessed via the General Self Efficacy (GSE) scale. Increases in GSE scores at 2-weeks would indicate beneficial effects on self efficacy.
Decision making efficacy | at baseline after 2 weeks of symptom monitoring
  Changes in Decision making efficacy scores as assessed via the Decision Self Efficacy (DSE) scale. Increases in DSE scores after 2-weeks would suggest benefical effects on medical decision making.
Health communication | at baseline after 2 weeks of symptom monitoring
  Changes in Health communication scores as assessed via the Willingness to Communicate about Health (WTCH) questionnaire. Increases in WTCH scores after 2-weeks would suggest benefical effects on health communication.
Health Anxiety | at baseline and after 2 weeks of symptom monitoring
  Changes in Health Anxiety scores as assessed via the Health Orientation Scale (HOS). Reductions in Health Anxiety after 2-weeks would suggest beneficial effects.
Health Consciousness | at baseline and after 2 weeks of symptom monitoring
  Changes in Health Consciousness scores as assessed via the HOS. Reductions in Health Consciousness scores after 2-weeks would suggest beneficial effects.
Coping preference | Measured at baseline to assess whether coping preference moderated symptom monitoring outcomes
  Monitoring/ Blunting Coping preference assessed via the Miller's Behavioural Style Scale (MBSS). The MBSS score can be used in analyses as a continuous variable, with individuals displaying more or less monitoring coping characteristics. Scores range from 0 (no monitoring characteristics) to 72 (high monitoring characteristics).
Trait neuroticism | Measured at baseline to assess whether trait neuroticism moderated symptom monitoring outcomes
  Trait neuroticism was assessed via the IPIP-NEO 10-item neuroticism subscale. This scale ranges from 10 (low trait neuroticism) to 50 (high trait neuroticism).

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Wales, Treforest, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews R, Hale G, John B, Lancastle D. Evaluating the Effects of Symptom Monitoring on Menopausal Health Outcomes: A Systematic Review and Meta-Analysis. Front Glob Womens Health. 2021 Dec 3;2:757706. doi: 10.3389/fgwh.2021.757706. eCollection 2021. PMID 34927137

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT05603234/Prot_SAP_ICF_000.pdf